CLINICAL TRIAL: NCT06004934
Title: An Open-Label, Phase 1 Study to Evaluate the Single-dose Pharmacokinetics of Avacopan (CCX168) in Male and Female Subjects With Mild or Moderate Hepatic Impairment
Brief Title: A Study to Evaluate the Pharmacokinetics of Avacopan (CCX168) in Participants With Mild or Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL013_168
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-07

CONDITIONS: Hepatic Impairment
Keywords: Liver disease; Anti-neutrophil cytoplasmic antibody-associated vasculitis; Complement C5a receptor (C5aR)
MeSH Terms: conditions — Liver Diseases; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — avacopan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment (defined using Child-Pugh Classification of the Severity of Liver Disease [C-P] criteria [C-P Class A, score of 5 to 6 points]) will receive a single oral dose of 30 mg avacopan on Day 1 in the fasted state.
  Interventions: Drug: Avacopan
- Group 2: Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment (defined using the C-P criteria [C-P Class B, score of 7 to 9 points]) will receive a single oral dose of 30 mg avacopan on Day 1 in the fasted state.
  Interventions: Drug: Avacopan
- Group 3: Healthy Control Group (Active Comparator): Participants with normal hepatic function (medically normal with no clinically significant illness or disease or abnormal physical examination findings, and with normal laboratory values at screening) will be demographically-matched to participants in Group 1 and Group 2, and will receive a single oral dose of 30 mg avacopan on Day 1 in the fasted state.
  Interventions: Drug: Avacopan

INTERVENTIONS:
Drug: Avacopan — Administered orally.
  Other Names: CCX168

SUMMARY:
The primary objective of this study will be to evaluate the pharmacokinetic properties of avacopan and its metabolite CCX168-M1 after a single oral dose of 30 mg avacopan in participants with mild or moderate hepatic impairment compared to matched healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board approved informed consent form is signed and dated prior to any study-related activities;
* Adult male or female participants, aged ≥18 to ≤75 years of age inclusive;
* Body mass index (BMI) ≥18.0 to ≤38.0 kg/m^2, inclusive, at screening;
* Female participants of childbearing potential or male participants with partners of childbearing potential may participate if adequate contraception is used during, and for at least 90 days after, any administration of study medication.

Inclusion Criteria Specific for Participants with Hepatic Impairment:

* Hepatic disease based on a documented history of hepatic insufficiency with features of cirrhosis and ability to classify hepatic disease as mild or moderate using C-P criteria;
* No acute episodes of illness related to hepatic insufficiency within 30 days prior to screening, and no significant change in disease status from screening to check-in (Day -1);
* On a stable medication regimen, defined as not starting any new prescription or non-prescription medications or significant changes in dose of such medications within 30 days prior to dosing of investigational drug on Day 1;
* Abnormal laboratory values must be clinically acceptable, as judged by the Investigator;
* Negative result of the human immunodeficiency virus (HIV) screen and the hepatitis B screen. Note hepatically impaired participants with chronic hepatitis C infection (duration > 6 months) are eligible for enrollment, if stable.

Inclusion criteria Specific for Healthy Participants:

* Participants must meet demographically-matched criteria to one of the participants enrolled in this study with moderate hepatic impairment based on sex, age (±10 years), and BMI (±20%);
* Medically normal with no clinically significant illness or disease and no significant abnormal findings at the baseline physical examination;
* Participant has normal (or abnormal and clinically insignificant) laboratory values at screening. A single test repeat at the discretion of the Investigator is allowed during the screening period to determine eligibility;
* Negative result from the HIV screen, the hepatitis B screen, and the hepatitis C screen.

Exclusion Criteria:

* Pregnant or breastfeeding;
* At least 7 days prior to check-in, and throughout the blood sample collection period, consumption of any food or any beverage containing grapefruit or grapefruit juice, Seville oranges, apple or orange juice, vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, cauliflower, Brussels sprouts, mustard greens) and charbroiled meats;
* Strenuous exercise within 4 days prior to check-in;
* Recent history of myopathy or muscle injury;
* Consumption of alcohol within 48 hours prior to check-in on Day -1 (as confirmed by alcohol test);
* A history or presence of any form of cancer within the 5 years prior to check-in, with the exception of excised basal cell or squamous cell carcinoma of the skin, or cervical carcinoma in situ or breast carcinoma in situ that has been excised or resected completely and is without evidence of local recurrence or metastasis;
* History or presence of unexplained syncope or family history of sudden death, or any medical condition or disease which, in the opinion of the Investigator, may place the participant at unacceptable risk for study participation;
* Donated or lost more than 350 mL of blood or blood products within 56 days prior to screening, or donated plasma within 7 days of dosing;
* Participant has any evidence of renal impairment; serum creatinine greater than 1.5 times the upper limit of normal at screening or check-in;
* Participant's urine tested positive at screening and/or check-in for any of the following (unless the positive drug screen in hepatic participants is due to prescription drug use and is approved by the investigator and the Sponsor's Medical Monitor): opioids, amphetamines and methamphetamines, cannabinoids, benzodiazepines, barbiturates, cocaine, cotinine (healthy participants only), methylenedioxymethamphetamine (MDMA or "ecstasy"), methadone, phencyclidine, tri-cyclic antidepressants, or alcohol;
* Currently taking a strong inducer of the cytochrome P450 3A4 (CYP3A4) enzyme, (e.g. carbamazepine, phenobarbital, phenytoin, rifampin, or St. John's wort) or use of a strong CYP3A4 inducer within 14 days prior to check-in and through discharge, unless deemed acceptable by the Investigator, Medical Monitor, and/or the Sponsor;
* Currently taking a strong inhibitor of the CYP3A4 enzyme, (e.g. boceprevir, clarithromycin, conivaptan, grapefruit juice, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, or voriconazoleor) or use of a strong CYP3A4 inhibitor within 14 days prior to check-in and through discharge, unless deemed acceptable by the Investigator, Medical Monitor, and/or the Sponsor;
* Participated in any clinical study of an investigational product within 30 days prior to dosing or within 5 half-lives after dosing;
* History within one year prior to check-in of illicit drug abuse;
* Significant infection or hospitalization within 28 days prior to check-in on Day -1.

Exclusion Criteria Specific for Participants with Hepatic Impairment:

* Currently on transplant list or history of portal shunts, recent variceal bleeds, or evidence of hepatorenal syndrome;
* History of prior liver transplant;
* For participants who are smokers, inability to restrict smoking to no more than 10 cigarettes per day from the screening visit until the last outpatient visit.

Exclusion Criteria Specific for Healthy Participants:

* Used a prescription and/or over-the-counter medication, with the exception of ibuprofen, hormonal contraceptives, and multi-vitamins, within 14 days prior to check-in; herbal supplements must be stopped 7 days prior to check-in;
* Participant's hemoglobin less than 11.5 g/dL for women or less than 13.0 g/dL for men, at screening or check-in, considered clinically significant by the investigator;
* Participant has any evidence of hepatic disease; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, or bilirubin greater than 1.5 times the upper limit of normal at screening or check-in;
* Participant's white blood cell count is below the lower limit of normal at screening or check-in, considered clinically significant by the investigator;
* Participant has used tobacco- or nicotine-containing products (e.g. cigarette, pipe, cigar, chewing, nicotine patch, or nicotine gum) within 6 months prior to check-in on Day -1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Avacopan | Up to Day 18
Cmax of CCX168-M1 | Up to Day 18
Time of Cmax (Tmax) of Avacopan | Up to Day 18
Tmax of CCX168-M1 | Up to Day 18
Terminal Phase Rate Constant of Avacopan | Up to Day 18
Terminal Phase Rate Constant of CCX168-M1 | Up to Day 18
Apparent Terminal Half-life (t1/2z) of Avacopan | Up to Day 18
t1/2z of CCX168-M1 | Up to Day 18
Apparent Oral Clearance (CL/F) of Avacopan | Up to Day 18
CL/F of CCX168-M1 | Up to Day 18
Apparent Volume of Distribution (Vz/F) of Avacopan | Up to Day 18
Vz/F of CCX168-M1 | Up to Day 18
Area Under the Plasma Concentration-time Curve (AUC) from Time 0 to Time t (time of last quantifiable plasma concentration) (AUClast) of Avacopan | Up to Day 18
AUClast of CCX168-M1 | Up to Day 18
AUC from Time 0 to Time 6 Hours Post-dose (AUC0-6h) of Avacopan | Up to Hour 6
AUC0-6h of CCX168-M1 | Up to Hour 6
AUC from Time 0 to Time 12 Hours Post-dose (AUC0-12h) of Avacopan | Up to Hour 12
AUC0-12h of CCX168-M1 | Up to Hour 12
AUC from Time 0 to Infinity (AUC0-inf) of Avacopan | Up to Day 18
AUC0-inf of CCX168-M1 | Up to Day 18

SECONDARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to Day 18

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Clinical Pharmacology of Miami, Inc., Hialeah, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Miao S, Suso P, Furst JA, Hudson MG, Trivedi A. Effect of Mild or Moderate Hepatic Impairment on the Pharmacokinetics of Avacopan, a Small-Molecule Complement C5a Receptor Antagonist, for the Treatment of Antineutrophil Cytoplasmic Autoantibody-Associated Vasculitis. Clin Pharmacol Drug Dev. 2024 Sep;13(9):1000-1010. doi: 10.1002/cpdd.1444. Epub 2024 Jul 11. PMID 38993026
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com